CLINICAL TRIAL: NCT04197661
Title: A Study Evaluating Pharmacokinetics, Pharmacodynamics and Safety of Intravenous Administration of HSK3486 Injectable Emulsion in Healthy Elderly Subjects
Brief Title: Safety and Pharmacokinetics/Pharmacodynamics of HSK3486 in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSK3486-108
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Healthy Elderly Subjects
Keywords: Healthy Elderly Subjects
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Elderly groupⅠ (Active Comparator): Elderly groupⅠ 65 years or older 0.2 mg/kg HSK3486
  Interventions: Drug: HSK3486
- Elderly group Ⅱ (Active Comparator): Elderly group Ⅱ 65 years or older 0.3 mg/kg HSK3486
  Interventions: Drug: HSK3486
- Elderly group Ⅲ (Active Comparator): Elderly group Ⅲ 65 years or older 0.4 mg/kg HSK3486
  Interventions: Drug: HSK3486
- Non-elderly group IV (Active Comparator): Non-elderly group IV 18 to 64 years 0.4 mg/kg HSK3486
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486 — Intravenously infuse 0.2 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Other Names: HSK3486 0.2 mg/kg
  Arms: Elderly groupⅠ
Drug: HSK3486 — Intravenously infuse 0.3 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Other Names: HSK3486 0.3 mg/kg
  Arms: Elderly group Ⅱ
Drug: HSK3486 — Intravenously infuse 0.4 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Other Names: HSK3486 0.4 mg/kg
  Arms: Elderly group Ⅲ
Drug: HSK3486 — Intravenously infuse 0.4 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Other Names: HSK3486 0.4 mg/kg
  Arms: Non-elderly group IV

SUMMARY:
It is a single-center, open-label, dose-finding, Phase I clinical study evaluating the pharmacokinetics, pharmacodynamics, and safety characteristics of HSK3486 in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and fully understand the content, procedure and possible adverse effects before the trial starts;
2. Able to complete the study in compliance with the requirements of the clinical trial protocol;
3. Subjects (including their partners) are willing to voluntarily adopt an effective measure of contraception starting from screening to 6 months after the last dose of the investigational drug. See the attachment for specific contraceptive measures;
4. Males and females with full capacity for civil conduct, aged ≥ 18 years old (aged between 18 and 64 years old for the non-elderly group and ≥ 65 years old for the elderly group (inclusive));
5. Females weighing ≥ 45 kg and males weighing ≥ 50 kg, and with a body mass index (BMI) of ≥ 18 and ≤ 30 kg/m2 (BMI = Weight (kg)/height2(m2))(inclusive);
6. For all subjects, the body temperature should be between 35.9-37.6 °C, respiratory rate between 12-20 breaths/min, and SpO2 when inhaling > 95%; in addition, for subjects in the non-elderly group, the blood pressure should be between 90-140/60-90 mmHg and heart rate between 60-99 bpm; for those in the elderly group, the blood pressure should be between 90-160/60-100 mmHg and heart rate between 50-100 bpm;

Exclusion Criteria:

1. Smoke more than 5 cigarettes per day on average within 3 months prior to screening;
2. Patient having contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
3. Known sensitivity to HSK3486 excipients (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate, and sodium hydroxide); or history of drug allergies (including other anesthetics), allergic diseases, or those with hyperactive immuneresponse(allergies to various drugs and foods);
4. History of drug abuse or any signs of long-term use of benzodiazepines (such as insomnia, anxiety, spasms) within 3 months prior to screening;
5. Acute diseases with clinical significance (determined by the investigator) within 2 weeks prior to screening, including GI diseases and infections (such as respiratory or CNS infections);
6. History or evidence of cardiovascular diseases prior to screening: Uncontrolled hypertension [SBP ≥ 170 mmHg and/or DBP ≥ 105 mmHg without antihypertensive treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment], postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medication, II-III degree atrioventricular block (excluding patients with pacemakers), or QTcF interval ≥ 450 ms (Fridericia's correction formula);
7. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | -30 minutes before administration until 24 hours post administration on day 1
  Cmax（a measure of the body's exposure to HSK3486）will be compared between non-elderly subjects and elderly subjects.
Area under the concentration-time curve（AUC） | -30 minutes before administration until 24 hours post administration on day 1
  AUC（a measure of the body's exposure to HSK3486）will be compared between non-elderly subjects and elderly subjects.

SECONDARY OUTCOMES:
MOAA/S(modified observer's assessment of alert /sedation) | -5 minutes before administration until 1 hours post administration on day 1
  modified observer's assessment of alert /sedation
Bispectral index(BIS) | -5 minutes before administration until 1 hours post administration on day 1
  Bispectral index
Tmax | -30 minutes before administration until 24 hours post administration on day 1
  time to peak observed
Total clearance | -30 minutes before administration until 24 hours post administration on day 1
  Total clearance
blood pressure（systolic, diastolic and mean arterial pressure） | from the screening to 2 days post-dose
  safety endpoits

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, PhD, Study Director — Phase I Clinical Trial Laboratory，The First Hospital of Jilin University
Locations (1):
- Phase I Clinical Trial Laboratory, The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qin L, Ren L, Wan S, Liu G, Luo X, Liu Z, Li F, Yu Y, Liu J, Wei Y. Design, Synthesis, and Evaluation of Novel 2,6-Disubstituted Phenol Derivatives as General Anesthetics. J Med Chem. 2017 May 11;60(9):3606-3617. doi: 10.1021/acs.jmedchem.7b00254. Epub 2017 Apr 28. PMID 28430430